CLINICAL TRIAL: NCT02314130
Title: No-commercial Enteral Diet for Patients in Home Nutritional Therapy: Effects on Anthropometric and Biochemical Indices
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Tania Morais, PhD, Federal University of São Paulo
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1732/08
Record Dates: First submitted 2013-03-18; First posted 2014-12-11 (Estimated); Last update posted 2014-12-11 (Estimated); Status verified 2013-03

CONDITIONS: Malnutrition
MeSH Terms: conditions — Malnutrition | interventions — Diet Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dietary therapy Standardized diet (Experimental): The study was constituted by sixty-six patients, thirty-three in each group. Patients on not industrialized enteral diet (standardized diet group) entered at random in the study and were matched by gender, age, socioeconomic status and medical diagnosis to patients using commercial diet (commercial group). The evaluation consisted of anthropometric measures of weight, height, arm circumference, triceps skin fold and biochemical índices at baseline and at the end of the intervention.
  Interventions: Dietary Supplement: Dietary therapy
- Dietary therapy Commercial diet group (No Intervention): The study was constituted by sixty-six patients, thirty-three in each group. Patients on not industrialized enteral diet (standardized diet group) entered at random in the study and were matched by gender, age, socioeconomic status and medical diagnosis to patients using commercial diet (commercial group). The evaluation consisted of anthropometric measures of weight, height, arm circumference, triceps skin fold and biochemical índices at baseline and at the end of the intervention.

INTERVENTIONS:
Dietary Supplement: Dietary therapy — A enteral diet formulation was developed to meet dietary requirements of adult patients. The formulation was standarized in household measures so that caregivers would prepare it and delivered it at the patients' home. Anthropometric measurements and blood samples were taken at baseline and at the end of the intervention which lasted four months.
  Arms: Dietary therapy Standardized diet

SUMMARY:
The objective is to evaluate the effect of no-commercial enteral diet for patients in home nutritional therapy in anthropometric and biochemical indices comparing to patients using commercial enteral diets.

ELIGIBILITY:
Inclusion Criteria:

* patients in home nutritional therapy receiving no-commercial enteral diets

Exclusion Criteria:

* baseline diseases others than neurological

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2009-05; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Recovery of malnourished patients (weight, height, arm circumference) | Two years
  weight, height, arm circumference

CONTACTS AND LOCATIONS:
Overall Officials: Tania Morais, PhD, Principal Investigator — Federal of University of Sao Paulo
Locations (1):
- Federal University of Sao Paulo, São Paulo, São Paulo, Brazil

REFERENCES:
- [Background] Santos VF, Morais TB. Nutritional quality and osmolality of home-made enteral diets, and follow-up of growth of severely disabled children receiving home enteral nutrition therapy. J Trop Pediatr. 2010 Apr;56(2):127-8. doi: 10.1093/tropej/fmp033. Epub 2009 May 19. PMID 19454554